CLINICAL TRIAL: NCT02167776
Title: Cluster-randomized Study of Church-Based Intervention to Promote Male Circumcision in Tanzania
Brief Title: From Obstacles to Opportunities for Male Circumcision in Tanzania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1107011800
Record Dates: First submitted 2014-06-17; First posted 2014-06-19 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Male Circumcision

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Church-based teaching (Experimental): Teaching about male circumcision provided to church leaders in addition to standard teaching available from Ministry of Health.
  Interventions: Behavioral: Church-based teaching
- No church-based teaching (No Intervention): Standard of care. Teaching about male circumcision provided by Ministry of Health.

INTERVENTIONS:
Behavioral: Church-based teaching — In villages that are randomized to receive the intervention, Christian church leaders of both genders and all denominations will be invited to attend an educational seminar about male circumcision. This seminar will last for one day in each intervention village, and will use a curriculum that the investigators' team developed in 2012 based on prior focus group work. Seminars will be conducted in Kiswahili (the national language) and co-taught by a Tanzanian pastor and a Tanzanian clinician who works with the male circumcision outreach campaign. Church leaders will be taught medical, historical, religious, tribal, and social aspects of male circumcision and given tools to lead their congregations in the understanding and practice of male circumcision.
  Arms: Church-based teaching

SUMMARY:
Male circumcision has been demonstrated by three randomized trials to be a highly effective method of HIV prevention, leading the World Health Organization to recommend its widespread implementation. The investigators' prior work in Tanzania has shown that the acceptability and uptake of male circumcision depends highly on religious beliefs. The investigators hypothesize that the uptake of male circumcision can be increased in villages in which male circumcision is offered in conjunction with church-based teaching and practice, compared with villages in which male circumcision is not promoted through churches.

The investigators will conduct a community randomized trial in rural Tanzania, where the government is systematically providing free male circumcision via campaigns in villages in which rates of circumcision are low. Prior to the start of the campaign, villages will be randomized to receive or not to receive church-based and culturally-informed promotion of male circumcision. All villages will receive the standard non-church-based health education that accompanies male circumcision campaigns.

The investigators will compare rates of male circumcision, both by self-report and by demographic data collected at the time of circumcision, among men and boys before and after the campaign in intervention villages with church involvement versus control villages without church involvement.

DETAILED DESCRIPTION:
The investigators will conduct a mixed-methods study that will include a community cluster randomized trial, followed by focus group discussions in both intervention and control villages after completion of the trial. This trial will be performed in 16 villages in conjunction with a voluntary medical male circumcision outreach campaign that is being offered by the Tanzanian Ministry of Health in the northwest of the country. The campaign brings a team of clinicians to perform free male circumcisions in 2-3 villages at a time. The campaign routinely provides male circumcision and voluntary HIV counseling and testing to between one hundred to two hundred men per day and typically remains in a village for 3-6 weeks until demand for circumcision decreases.

The unit of randomization in the cluster randomized trial will be the village. The investigators will work in partnership with the male circumcision outreach campaign to identify eligible village pairs that are located within 60 kilometers of one another and will be targeted by the male circumcision outreach campaign at the same time. The investigators believe that the geographic proximity of the paired villages and the start date of the male circumcision outreach campaign in the village will be the two most important factors affecting uptake of male circumcision in the villages. The geographic proximity is important for the assumption that baseline rates of male circumcision and other village characteristics are likely similar. The start date of the campaign is important because: (1) uptake of male circumcision is likely to be higher during the dry season, when there is less farming work for men to do, and (2) the investigators predict that uptake of male circumcision may increase over time as more and more men are circumcised in the Mwanza region and it increasingly becomes a societal norm.

The investigators will restrict our inclusion criteria to rural villages that have clear boundaries so that the male population is stable without influx as would be common in an urban area. In these rural regions, dirt roads and poor infrastructure lead to minimal contact between villages so it is predicted that little information will be shared between intervention and control villages.

Both intervention and control villages will receive the standard community outreach events to promote male circumcision that are provided by the Tanzanian Ministry of Health during their male circumcision outreach campaign. This may include community meetings, public education sessions by health care workers, drama, broadcast announcements by cars with megaphones, and distribution of health informational brochures. However, the standard education does not work specifically with religious leaders. Among the members of the male circumcision outreach team, only one clinician, who will provide medical teaching at the educational seminar for religious leaders, will be aware of a village's assignment as an intervention or control group.

The additional intervention that will be given to villages that are randomized to receive the intervention will be a one-day educational seminar for church leaders of that village. The seminar will focus on male circumcision and will address religious, cultural, and health implications of this practice. It will also provide teaching and tools for church leaders to use in discussing male circumcision with their congregations.

After the completion of the male circumcision outreach campaign in a village, our study team will enroll individual church leaders. Leaders from both intervention and control villages will participate in separate groups and will be led in a discussion of their perceptions of male circumcision. Church leaders, who will be invited from a variety of denominational backgrounds, will provide written informed consent for participation in the focus group discussions.

ELIGIBILITY:
Inclusion Criteria:

* Villages in which male circumcision is being offered by the Tanzanian Ministry of Health free of charge
* Village leader provides permission for study participation

Exclusion Criteria:

-

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
rate of uptake of male circumcision | 9 months

SECONDARY OUTCOMES:
qualitative data from church attenders in intervention and control villages | 9 months

OTHER OUTCOMES:
age-specific rates of male circumcision uptake | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Downs, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Bugando Medical Centre and catchment area, Mwanza, Tanzania

IPD SHARING:
Plan to Share IPD: Undecided